CLINICAL TRIAL: NCT01472887
Title: An Open Label Non-Randomized Phase 2 Study Evaluating SAR3419, an Anti-CD19 Antibody - Maytansine Conjugate, Administered as Single Agent by Intravenous Infusion to Patients With Relapsed or Refractory CD19+ Diffuse Large B-Cell Lymphoma
Brief Title: SAR3419 as Single Agent in Relapsed-Refractory Diffuse Large B-Cell Lymphoma (DLBCL) Patients
Acronym: STARLYTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD10248; 2011-003657-26; U1111-1115-3349 (Other: UTN)
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — coltuximab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR3419 (Experimental): All patients will receive SAR3419 until evidence of disease progression, unacceptable toxicity, or other reasons for therapy discontinuation
  Interventions: Drug: SAR3419

INTERVENTIONS:
Drug: SAR3419 — Pharmaceutical form:concentrate for solution for infusion
  Route of administration: intravenous

SUMMARY:
Primary Objective:

Participants achieving an Objective Response Rate

Secondary Objective:

* Progression Free Survival
* Overall Survival
* Response Duration
* Safety

DETAILED DESCRIPTION:
The screening period = up to 4 weeks prior to SAR3419 administration

The treatment period = from the day of first administration of SAR3419 until the End-Of-Treatment visit. All patients will receive SAR3419 until evidence of disease progression, unacceptable toxicity or other reasons for therapy discontinuation - After therapy discontinuation all patients will enter a safety follow-up period of 42 days starting from the day of administration of the last dose of SAR3419 and ending with the End Of Treatment visit.

All patients, regardless whether they have progressed or not, will be followed until death or end of study to evaluate survival for at least 18 months.

ELIGIBILITY:
Inclusion criteria:

* Histological diagnosis of Diffuse Large B Cell Lymphoma (de novo or transformed) expressing CD19 by immunohistochemistry or flow cytometry analysis (>30% positivity), based on recent (less than 6 months) or new biopsy.
* At least 1 prior specific therapeutic regimen, one of which should have included rituximab (patients previously eligible for transplantation: the salvage treatment followed by intensification and Autologous Stem Cell Transplant (ASCT) will be considered one regimen).
* Relapsed disease after standard 1st line therapy for aggressive lymphoma - not eligible for high dose chemotherapy with stem cell support. Relapsed or refractory disease after two lines of therapy one of which could have included Autologous Stem Cell Transplant (ASCT). Relapsed disease is defined as progression after a disease free interval of at least 6 months after completion of last therapy. Refractory is defined as progression of disease during prior therapy or within 6 months from its completion.
* Available paraffin-embedded tissue should have been collected no longer than 6 months prior to first administration of SAR3419. Cryo-preserved tissue cannot be used. If archival material is not available, a Fine Needle Aspiration (FNA) must be obtained.

Exclusion criteria:

* Primary refractory patients
* Patients with primary mediastinal DLBCL

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of participants achieving an Objective Response Rate | 18 months

SECONDARY OUTCOMES:
Number of participants with Adverse Events | Up to 1 year
Response duration - Time | Up to 18 months after the first infusion of the last patient
Progression Free Survival - Time | Up to 18 months after the first infusion of the last patient
Overall Survival - Time | Up to 18 months after the first infusion of the last patient

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (28):
- United States (3):
  - Investigational Site Number 840001, Denver, Colorado
  - Investigational Site Number 840003, Augusta, Georgia
  - Investigational Site Number 840005, Boise, Idaho
- Belgium (2):
  - Investigational Site Number 056002, Ghent
  - Investigational Site Number 056001, Leuven
- Czechia (3):
  - Investigational Site Number 203002, Brno
  - Investigational Site Number 203003, Prague
  - Investigational Site Number 203001, Prague
- Israel (2):
  - Investigational Site Number 376003, Jerusalem
  - Investigational Site Number 376002, Tel Litwinsky
- Italy (7):
  - Investigational Site Number 380002, Bergamo
  - Investigational Site Number 380004, Bologna
  - Investigational Site Number 380008, Mestre
  - Investigational Site Number 380001, Milan
  - Investigational Site Number 380007, Modena
  - Investigational Site Number 380003, Palermo
  - Investigational Site Number 380006, Pavia
- Poland (3):
  - Investigational Site Number 616003, Brzozów
  - Investigational Site Number 616002, Kielce
  - Investigational Site Number 616001, Warsaw
- Spain (4):
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724004, Barcelona
  - Investigational Site Number 724001, Madrid
  - Investigational Site Number 724003, Valencia
- Turkey (Türkiye) (2):
  - Investigational Site Number 792003, Izmir
  - Investigational Site Number 792001, Izmir
- United Kingdom (2):
  - Investigational Site Number 826001, Leicester
  - Investigational Site Number 826002, Manchester

REFERENCES:
- [Derived] Trneny M, Verhoef G, Dyer MJ, Ben Yehuda D, Patti C, Canales M, Lopez A, Awan FT, Montgomery PG, Janikova A, Barbui AM, Sulek K, Terol MJ, Radford J, Guidetti A, Di Nicola M, Siraudin L, Hatteville L, Schwab S, Oprea C, Gianni AM. A phase II multicenter study of the anti-CD19 antibody drug conjugate coltuximab ravtansine (SAR3419) in patients with relapsed or refractory diffuse large B-cell lymphoma previously treated with rituximab-based immunotherapy. Haematologica. 2018 Aug;103(8):1351-1358. doi: 10.3324/haematol.2017.168401. Epub 2018 May 10. PMID 29748443